CLINICAL TRIAL: NCT05546593
Title: Prevalence of Abnormalities in Ultrasonography of Joint and Tendons in Patients With Gout
Acronym: EchoGoutte
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220681; 2022-A01121-42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Gout
Keywords: Gout; Ultrasound; Microcrystal disease
MeSH Terms: conditions — Gout; Elephantiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gout is the most frequent inflammatory arthritis in men after 40 years, with a prevalence of 0.9% in France. This disease is characterized by deposits of sodium urate crystals in joints, tendons and soft tissues, which can be detected by ultrasound examination. To date, there was no study assessing inflammatory, structural and deposit lesions due to gout in joints and tendons, since the standardization of ultrasound definitions of gout by the OMERACT (Outcome Measures in Rheumatology) in 2015. The objective of this study is t estimate the prevalence and severity of ultrasound inflammatory lesions (synovitis, tenosynovitis, soft tissues abnormalities), structural lesions (osteophytes, erosions) and abnormalities due to sodium urate deposits (double contour, aggregates, tophi) in patients with gout.

DETAILED DESCRIPTION:
Gout is the most frequent inflammatory arthritis in men after 40 years, with a prevalence of 0.9% in France. This disease is characterized by deposits of sodium urate crystals in joints, tendons and soft tissues, which can be detected by ultrasound examination. To date, there was no study assessing inflammatory, structural and deposit lesions due to gout in joints and tendons, since the standardization of ultrasound definitions of gout by the OMERACT (Outcome Measures in Rheumatology) in 2015. The objective of this study is t estimate the prevalence and severity of ultrasound inflammatory lesions (synovitis, tenosynovitis, soft tissues abnormalities), structural lesions (osteophytes, erosions) and abnormalities due to sodium urate deposits (double contour, aggregates, tophi) in patients with gout. This is a transversal bicentric study, including patients who consulted for gout in the Rheumatology and Internal Medicine department of Ambroise Paré Hospital. Inclusion criteria were adult patients with a diagnosis of gout according to ACR/EULAR 2015 criteria and able to give informed consent. Exclusion criteria were the presence of other chronic inflammatory rheumatic diseases and patients without French social insurance. Patients had clinical and ultrasound examination, realized by two physicians blinded from each other.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were adult patients with a diagnosis of gout according to ACR/EULAR 2015 criteria and able to give informed consent. Exclusion criteria were the presence of other chronic inflammatory rheumatic diseases and patients without French social insurance.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in Rheumatology or Internal Medicine Departments of Ambroise Paré hospital-APHP.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Ultrasound lesion of gout as defined by OMERACT (Outcome Measures in Rheumatology) | at baseline
  double contour, agreggates, tophi, erosions, synovitis, tenosynovitis and osteophytes

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Antonietta D'AGOSTINO, MD, PhD, Principal Investigator — Rhumatology department, Ambroise Paré hospital - APHP
Locations (1):
- Rhumatology department, Ambroise Paré hospital - APHP, Boulogne-Billancourt, APHP, France